CLINICAL TRIAL: NCT03782584
Title: Efficiency of Modified Pilates Exercises in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gonca Şahiner Pıçak, associate professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEU.HSI.MSc-2015970022
Record Dates: First submitted 2018-03-19; First posted 2018-12-20 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2018-12

CONDITIONS: Neck Pain
Keywords: exercise; pilates; modified pilates; chronic neck pain
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Pilates Exercise Group (Experimental): they will be involved in a modified pilates exercise training for a total of 6 weeks a day, 2 days a week.
  Interventions: Other: modified pilates exercise
- Control Group (Other): they will be given daily life advises to prevent neck pain
  Interventions: Other: daily life advises

INTERVENTIONS:
Other: modified pilates exercise — modified exercises from original pilates exercises.
  Other Names: daily routine advises
  Arms: Modified Pilates Exercise Group
Other: daily life advises — they will be given daily life advises to prevent neck pain
  Arms: Control Group

SUMMARY:
The aim of this study is to investigate the effects of modified pilates exercises on neck pain, deep neck flexor muscles edurance, joint position sense and functionality in patients with chronic neck pain.

DETAILED DESCRIPTION:
50 individuals with Chronic Neck Pain not working will be included to our study. We will evaluate pain (with visual analog scale), deep neck flexors' endurance (with cranio-cervical flexure test using the pressure stabilizing feedback device), cervical range of motion and cervical proprioception (wit cervical range of motion device). Besides we will conduct a questionnaire (neck disability index) to get further knowledge about their functionality. Participants will be randomly allocated 2 groups consisting of 25 participants and these 2 groups will receive different interventions. Modified Pilates Exercise Group (MPEG) will be involved in a modified pilates exercise training for a total of 6 weeks a day, 2 days a week in the presence of a physiotherapist. The Control Group (KG) will receive daily routine advises to prevent neck pain and they will be asked about to apply these advises and not to make other changes in their life. The evaluations will be repeated and analyzed 2 times, pre-treatment and 6 weeks after treatment , and the effectiveness of the modified pilates exercises will be examined in the chronic neck pain. Our hypothesis is ''Modified pilates exercises have a positive effect on neck pain, range of motion, deep neck flexor muscles, joint position sense and function in patients with chronic neck pain.''

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain more than 3 months
* No physical therapy in last year
* No background with pilates exercises
* Being able to understand Turkish, treatment and evaluations.
* Being able to complete all the evaluations and treatment

Exclusion Criteria:

* Fracture or surgery background with shoulder, cervical area or other extremities.
* Any systemic musculoskeletal diseases
* Existing chest deformities or scoliosis
* Cervical hernia, neuropathy or whiplash.
* Pregnancy
* Having pain above 7 in VAS
* Any other pain that could prevent people from doing exercises

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Pain Evaluation | 6 weeks
  This test will be measured by Visual Analog Scale (VAS) score. VAS has 10-centimeter line corresponding to the amount of pain they experienced. "0" means "no pain" and "10" means "pain as bad as possible".
Neck Disability Index | 6 weeks
  Neck disability index is a survey that has 10 different sections including Pain intensity, personal care, weight lifting, reading, headache, concentration, work, driving, sleeping and resting activitie.
Posture Evaluation | 6 weeks
  Sagital plan photographs of the people will be taken and head and shoulder posture will be evaluated.
Neck Range Of Motion | 6 weeks
  Range of motion will be measured by cervical range of motion device (CROM device)
Deep Neck Flexor Endurance | 6 weeks
  Score of cranio-cervical flexion test will be measured by Stabilizer Pressure Biofeedback Unit.
Neck Position Sense | 6 weeks
  Joint position error of 6-direction (flexion, extension, right-left lateral flexion and right-left rotation) will be measured by cervical range of motion device (CROM device).

CONTACTS AND LOCATIONS:
Overall Officials: sevgi sevi yeşilyaprak, PHD, Principal Investigator — 9 eylül university
Locations (1):
- Izmir University of Economics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sahiner Picak G, Yesilyaprak SS. Effects of clinical pilates exercises in patients with chronic nonspecific neck pain: a randomized clinical trial. Ir J Med Sci. 2023 Jun;192(3):1205-1214. doi: 10.1007/s11845-022-03101-y. Epub 2022 Jul 20. PMID 35857170